CLINICAL TRIAL: NCT03359356
Title: Defining Reversal of Alopecia Areata (AA) Phenotype With Dupilumab in Patients With and Without Associated Atopic Dermatitis (AD)
Brief Title: Treatment of Alopecia Areata (AA) With Dupilumab in Patients With and Without Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Rockefeller University (Other); Regeneron Pharmaceuticals (Industry); Sanofi (Industry)
Responsible Party: Principal Investigator, Emma Guttman, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 17-1084
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Alopecia Areata
Keywords: alopecia; alopecia areata; alopecia universalis; alopecia totalis; dupixent; dupilumab
MeSH Terms: conditions — Alopecia Areata; Alopecia; Alopecia universalis | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dupilumab (Experimental): An initial dupilumab dose of 600 mg (two 300 mg subcutaneous injections), followed by dupilumab 300 mg given every week
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): Matching placebo in prefilled syringes identical to the dupilumab syringes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — A total of 24 doses
  Other Names: Dupixent
  Arms: Dupilumab
Drug: Placebo — A total of 24 doses
  Other Names: matching placebo
  Arms: Placebo

SUMMARY:
Alopecia areata is a medical condition, in which the hair falls out in patches. The hair can fall out on the scalp or elsewhere on the face and body. Alopecia areata is an autoimmune skin disease, which means that the immune system is recognizing the hair follicles as foreign and attacking them, causing round patches of hair loss. It can progress to total scalp hair loss (alopecia totalis) or complete body hair loss (alopecia universalis). The scalp is the most commonly affected area, but the beard or any hair-bearing site can be affected alone or together with the scalp. Alopecia areata occurs in males and females of all ages, and is a highly unpredictable condition that tends to recur. Alopecia areata can cause significant distress to both patients and their families. In this study, the aim is to assess the effects of dupilumab in patients with alopecia areata.

DETAILED DESCRIPTION:
The purpose of this study is to assess whether dupilumab can be a helpful treatment for alopecia areata.

This is a randomized, double-blind, placebo-controlled pilot study of a total of 54 subjects with moderate to severe alopecia areata involving 30-100% of the scalp. The researchers expect one third of these subjects to have concomitant alopecia areata (AA) and atopic dermatitis (AD).

The researchers' experience in AD, and past experience in psoriasis showed that biomarker studies in skin tissues are critical to the understanding of key pathogenic pathways that are upregulated in each disease and how well they are suppressed with effective treatment. These mechanistic studies coupled with clinical trials are key in the disease to shed light on important disease mechanisms, and to explain which molecules are suppressed by each therapeutic target. Data shows that IL-13 is significantly upregulated in both AD and AA lesions compared to nonlesional skin. It is very important to associate the clinical responses with suppression of this cytokine and related molecules as well as other pathway cytokines in skin tissues. Both the whole genomic profiling and individual molecular and cellular markers are very important in order to understand how well anti-IL-13 will change/suppress AA-associated pathways and compare with those that will be suppressed in AD.

Since this study is designed to gain basic knowledge rather than to yield information directly related to patient care, the results are not entered in the participants' medical records. If, at a later date, correlations of in-vitro tests and the patients' clinical situation suggest that the results do bear on the patients' health, an amended protocol will be submitted to the IRB so that results can be made available to the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are at least 18 years old at the time of informed consent.
* Subject is able to understand and voluntarily sign an informed consent document prior to participation
* Subject is able to adhere to the study visit schedule and other protocol requirements.
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product (IP), FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

  1. Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR
  2. Option 2: Male or female condom (latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]); PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.
* If subject is a female of non-childbearing potential, she must have documented history of infertility, be in a menopausal state for one year, or had a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy.
* Subject has a history of at least 6 months of moderate to severe AA (≥ 30% scalp involvement) as measured using the SALT score; OR subject has ≥ 95% loss of scalp hair for enrollment as AA totalis (AT) or universalis (AU) subtypes.

  1. AT and AU will be limited to 50% of the total number of subjects enrolled.
  2. One-third of subjects must have active AD skin or a concomitant history of AD at the time of the Screening and Baseline visits.
* Subject has a negative Tuberculin purified protein derivative (PPD) or QuantiFERON TB-Gold test (QFT) prior to baseline. Subjects with a positive or indeterminable PPD or QFT result must have a documented negative workup for tuberculosis and/or completed standard tuberculosis therapy.
* Subjects must meet the following laboratory criteria:

  1. White blood cell count ≥ 3000/mm3 (≥ 3.0 x 109/L) and < 14,000/mm3 (≤ 14 x 109/L).
  2. Platelet count ≥ 100,000/μL (≥ 100 x 109/L).
  3. Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L).
  4. AST (SGOT) and ALT (SGPT) ≤ 2 x upper limit of normal (ULN). If the initial test shows ALT or AST > 2 times the ULN, one repeat test is allowed during the Screening Phase.
  5. Total bilirubin ≤ 2 mg/dL (34 μmol/L). If the initial test shows total bilirubin > 2 mg/dL (34 μmol/L), one repeat test is allowed during the Screening Phase.
  6. Hemoglobin ≥ 10 g/dL (≥ 6.2 mmol/L).
* Subject is judged to be in otherwise good overall health following a detailed medical and medication history, physical examination, and laboratory testing.

Exclusion Criteria:

* Subject is pregnant or breastfeeding.
* Subject's cause of hair loss is indeterminable and/or they have concomitant causes of alopecia, such traction, cicatricial, pregnancy-related, drug-induced, telogen effluvium, or advanced androgenetic alopecia (i.e. Ludwig Type III or Norwood-Hamilton Stage ≥ V).
* Subject has a history of AA with no evidence of hair regrowth for ≥ 10 years since their last episode of hair loss.
* Subject has an active bacterial, viral, or helminth parasitic infections; OR a history of ongoing, recurrent severe infections requiring systemic antibiotics
* Subject with a known or suspected underlying immunodeficiency or immune-compromised state as determined by the investigator.
* Subject has a concurrent or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, intestinal, metabolic, endocrine, pulmonary, cardiovascular, or neurological disease.
* Active hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or positive HIV serology at the time of screening for subjects determined by the investigators to be at high-risk for this disease.
* Subject has a suspected or active lymphoproliferative disorder or malignancy; OR a history of malignancy within 5 years before the Baseline assessment, except for completely treated in situ non-melanoma skin and cervical cancers without evidence of metastasis.
* Subject has received a live attenuated vaccine ≤ 30 days prior to study randomization.
* Subject has any uncertain or clinically significant laboratory abnormalities that may affect interpretation of study data or endpoints.
* Subject has any other medical or psychological condition that, in the opinion of the investigator, may present additional unreasonable risks as a result of their participation in the study and/or interfere with clinic visits and necessary study assessments.
* History of adverse systemic or allergic reactions to any component of the study drug.
* Severe, untreated asthma or a history of life-threatening asthma exacerbations while on appropriate anti-asthmatic mediations.
* Use of systemic immunosuppressive medications, including, but not limited to, cyclosporine, systemic or intralesional corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, tacrolimus, or ultraviolet (UV) phototherapy with/without Psoralen Ultraviolet A (PUVA) therapy within 4 weeks prior to randomization.
* Use of an oral JAK inhibitor (tofacitinib, ruxolitinib) within 12 weeks prior to the Baseline visit.
* Subject has used topical corticosteroids, and/or tacrolimus, and/or pimecrolimus within 1 week before the Baseline visit.
* Subject has been previously treated with dupilumab.
* Subject currently uses or plans to use anti-retroviral therapy at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD,PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Rockefeller University Laboratory for Investigative Dermatology, New York, New York

IPD SHARING:
Plan to Share IPD: No
Since this study is designed to gain basic knowledge rather than to yield information directly related to patient care, the results are not entered in the participants' medical records. If, at a later date, correlations of in-vitro tests and the patients' clinical situation suggest that the results do bear on the patients' health, an amended protocol will be submitted to the IRB so that results can be made available to the medical record.

REFERENCES:
- [Derived] Guttman-Yassky E, Renert-Yuval Y, Bares J, Chima M, Hawkes JE, Gilleaudeau P, Sullivan-Whalen M, Singer GK, Garcet S, Pavel AB, Lebwohl MG, Krueger JG. Phase 2a randomized clinical trial of dupilumab (anti-IL-4Ralpha) for alopecia areata patients. Allergy. 2022 Mar;77(3):897-906. doi: 10.1111/all.15071. Epub 2021 Sep 6. PMID 34460948

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Dupilumab: Placebo given Weeks 0-24, then Dupilumab given Weeks 24-48
  Matching placebo in prefilled syringes identical to the dupilumab syringes. After 24 weeks of Placebo, an initial dose of 600 mg Dupilumab (two 300 mg subcutaneous injections), followed by open-label period in which 300 mg given every other week. A total of 24 Dupilumab doses.
- Dupilumab: An initial dose of 600 mg (two 300 mg subcutaneous injections), followed by 300 mg given every other week. A total of 48 Dupilumab doses will be given throughout the clinical trial, including 24 weeks during a randomized period and 24 weeks during an open label period.
Period: Overall Study
Arm/Group | Placebo Then Dupilumab | Dupilumab
Started | 20 | 40
Completed | 20 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Then Dupilumab: Matching placebo in prefilled syringes identical to the dupilumab syringes. After 24 weeks of Placebo, an initial dose of 600 mg Dupilumab (two 300 mg subcutaneous injections), followed by an open-label period in which 300 mg given every other week. A total of 24 Dupilumab doses.
- Total: Total of all reporting groups
Arm/Group | Placebo Then Dupilumab | Dupilumab | Total
Number analyzed (Participants) | 20 | 40 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (14.4) | 41.6 (13.8) | 43 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 30 | 43
  Male | 7 | 10 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 31 | 46
  African American | 2 | 3 | 5
  Asian | 2 | 6 | 8
  Other | 1 | 0 | 1
Duration since last hair regrowth [Mean (Standard Deviation); unit: years] | 3.5 (3) | 3.8 (2.9) | 3.6 (3)
Severity of alopecia tool (SALT) [Mean (Standard Deviation); unit: units on a scale] — SALT score 0-100 with lower score indicating better health outcomes
  units on a scale | 75.4 (26.1) | 70.5 (27.6) | 72.1 (27)
Patients with SALT>75 [Count of Participants; unit: Participants] | 12 | 20 | 32
Patients with SALT<75 [Count of Participants; unit: Participants] | 8 | 20 | 28
Patients with Alopecia Totalis/Universalis [Count of Participants; unit: Participants] | 8 | 13 | 21
Alopecia Areata Symptom Impact Scale (AASIS) score [Mean (Standard Deviation); unit: units on a scale] — AASIS score 0-130 with lower score indicating better health outcomes
  units on a scale | 56.1 (32.86) | 48.42 (30.27) | 50.9 (31.33)
Alopecia Areata Quality of Life (AA-QoL) score [Mean (Standard Deviation); unit: units on a scale] — AA-QoL score 0-100 with higher score indicating better health outcomes
  units on a scale | 51.75 (13.88) | 49.49 (12.56) | 50.25 (13.1)
Eyelash assessment [Count of Participants; unit: Participants] — 0 (none) to 4 (prominent) scale to stage hair status in eyelashes. Population: One participant had missing eyelash data at baseline because of artificial eyelashes (glued on her real eyelashes)
  Participants
    Very prominent: number analyzed (Participants) | 19 | 40 | 59
    Very prominent | 6 | 12 | 18
    Prominent: number analyzed (Participants) | 19 | 40 | 59
    Prominent | 2 | 6 | 8
    Moderate: number analyzed (Participants) | 19 | 40 | 59
    Moderate | 1 | 4 | 5
    Minimal: number analyzed (Participants) | 19 | 40 | 59
    Minimal | 6 | 9 | 15
    None: number analyzed (Participants) | 19 | 40 | 59
    None | 4 | 9 | 13
Eyebrow assessment [Count of Participants; unit: Participants] — 0 (none) to 4 (prominent) scale to stage hair status in eyelashes.
  Participants
    Very prominent | 6 | 10 | 16
    Prominent | 0 | 5 | 5
    Moderate | 2 | 6 | 8
    Minimal | 8 | 9 | 17
    None | 4 | 10 | 14
Patients with atopic dermatitis (AD) history [Count of Participants; unit: Participants] | 6 | 17 | 23
Patients with active AD [Count of Participants; unit: Participants] | 2 | 5 | 7
Eczema area and severity index (EASI) score [Mean (Standard Deviation); unit: units on a scale] — The EASI index assigns proportionate values to 4 body regions. Each region is assigned a score of 0 to 3, indicating none, mild, moderate, and severe clinical expression. The percentage of area involved is also assigned an eruption proportional score from 0 to 6. The total body score for each body region is obtained by multiplying the sum of the severity scores by the area score, then multiplying the result by the constant weighted value assigned to that body region. The sum of these scores gives the EASI total from 0-72, with higher score indicating more severity.
  units on a scale | 27.4 (11.0) | 13.58 (5.68) | 17.53 (9.83)
Patients with family history of atopy [Count of Participants; unit: Participants] | 9 | 18 | 27
IgE [Mean (Standard Deviation); unit: IU/ml] | 342.5 (826.7) | 525.8 (1211.3) | 464.7 (1094)
Patients with IgE≥200 [Count of Participants; unit: Participants] | 5 | 13 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Severity of Alopecia Tool (SALT) Score at Week 24
Description: The SALT is a validated instrument for measuring the amount of scalp hair loss at a single point in time The SALT is a validated instrument for measuring the amount of scalp hair loss at a single point in time SALT - Scalp divided into four areas: vertex (40% of scalp surface area), right profile (18% of scalp surface area), left profile (18% of scalp surface area), and posterior scalp (24% of scalp surface area). Percentage of hair loss in these areas is multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all areas. SALT scores range from 0 (no hair loss) to 100 (complete scalp hair loss) with lower score indicating better health outcomes/less hair loss. Primary Outcome is baseline minus Week 24 value.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Then Dupilumab | Dupilumab
Number analyzed (Participants) | 20 | 40
score on a scale | -6.3 (4.2) | 2.3 (3)

2. Secondary Outcome: Change From Week 24 in the SALT Score at Week 48
Description: SALT - Scalp divided into four areas: vertex (40% of scalp surface area), right profile (18% of scalp surface area), left profile (18% of scalp surface area), and posterior scalp (24% of scalp surface area). Percentage of hair loss in these areas is multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all areas. Week 24 minus week 48 value.
Time Frame: Week 24 and 48 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Then Dupilumab | Dupilumab
Number analyzed (Participants) | 20 | 40
score on a scale | -6.3 (4.2) | 2.3 (3)

3. Secondary Outcome: Change From Baseline in the SALT Score at Week 48
Description: Change in SALT score at Week 48 compared to Baseline. SALT - Scalp divided into four areas: vertex (40% of scalp surface area), right profile (18% of scalp surface area), left profile (18% of scalp surface area), and posterior scalp (24% of scalp surface area). Percentage of hair loss in these areas is multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all areas. SALT scores range from 0 (no hair loss) to 100 (complete scalp hair loss) with lower score indicating better health outcomes/less hair loss. Baseline minus week 48 value.
Time Frame: Baseline and 48 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Then Dupilumab | Dupilumab
Number analyzed (Participants) | 20 | 40
score on a scale | -6.3 (4.2) | 2.3 (3)

4. Secondary Outcome: Number of Patients Achieving at Least 50% Improvement in Severity of Alopecia Tool (SALT) Score (SALT-50) at Weeks 24 and 48 Compared to Baseline
Description: Number of subjects achieving SALT-50 score at Weeks 24 and 48 compared to Baseline. SALT - Scalp divided into four areas: vertex (40% of scalp surface area), right profile (18% of scalp surface area), left profile (18% of scalp surface area), and posterior scalp (24% of scalp surface area). Percentage of hair loss in these areas is multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss SALT scores range from 0 (no hair loss) to 100 (complete scalp hair loss) with lower score indicating better health outcomes/less hair loss.in all areas.
Time Frame: weeks 24 and 48
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Then Dupilumab: Matching placebo in prefilled syringes identical to the dupilumab syringes. After 24 weeks, an initial dose of 600 mg (two 300 mg subcutaneous injections), followed by 300 mg given every other week. A total of 24 doses.
- Dupilumab: An initial dose of 600 mg (two 300 mg subcutaneous injections), followed by 300 mg given every other week, A total of 24 doses
Arm/Group | Placebo Then Dupilumab | Dupilumab
Number analyzed (Participants) | 20 | 40
Participants
  Week 24 | 0 | 4
  Week 48 | 3 | 9

5. Secondary Outcome: Number of Patients Achieving at Least 75% Improvement in SALT-75 at Weeks 24 and 48
Description: Number of patients with Severity of Alopecia Tool (SALT) Score (SALT-75) (> or equal to 75% improvement in SALT score) at Weeks 24 compared to Baseline. SALT - Scalp divided into four areas: vertex (40% of scalp surface area), right profile (18% of scalp surface area), left profile (18% of scalp surface area), and posterior scalp (24% of scalp surface area). Percentage of hair loss in these areas is multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all areas. SALT scores range from 0 (no hair loss) to 100 (complete scalp hair loss) with lower score indicating better health outcomes/less hair loss.
Time Frame: Weeks 24 and 48
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Then Dupilumab | Dupilumab
Number analyzed (Participants) | 20 | 40
Participants
  Week 24 | 0 | 2
  Week 48 | 1 | 6

6. Secondary Outcome: Number of Patients Achieving at Least 90% Improvement in Severity of Alopecia Tool (SALT) Score (SALT-90) at Weeks 24 and 48
Description: The number of patients achieving at least 90% improvement in Severity of Alopecia Tool (SALT) score (SALT-90) at Weeks 24, 48 compared to Baseline
Time Frame: Weeks 24 and 48
Measure: Count of Participants; unit: Participants
Groups:
- Dupilumab: An initial dose of 600 mg (two 300 mg subcutaneous An initial dose of 600 mg (two 300 mg subcutaneous injections), followed by 300 mg given every other week. A total of 48 Dupilumab doses will be given throughout the clinical trial, including 24 weeks during a randomized period and 24 weeks during an open label period.), followed by 300 mg given every other week, A total of 24 doses
Arm/Group | Placebo Then Dupilumab | Dupilumab
Number analyzed (Participants) | 20 | 40
Participants
  Week 24 | 0 | 1
  Week 48 | 1 | 4

7. Secondary Outcome: Change in Alopecia Areata Symptom Impact Scale (AASIS)
Description: Change in AASIS at Weeks 24 and 48 compared to Baseline. AASIS is a 13-item instrument, each item scored from 0 to 10 where higher scores correspond to worse symptom impact, full range from 0 to 130.
Time Frame: Weeks 24 and 48
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Matching placebo in prefilled syringes identical to the dupilumab syringes. A total of 24 doses
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 20 | 40
score on a scale
  Week 24 | 10.25 (20.29) | 0.64 (22.27)
  Week 48 | 22.6 (35.42) | 8.13 (27.65)

8. Secondary Outcome: Change in Alopecia Areata Quality of Life Questionnaire
Description: Change in the Alopecia Areata Quality of Life questionnaire (AA-QoL) at Weeks 24 and 48 compared to baseline. AAQoL is a 21-item instrument scored from 0 (poor) to 100 (good).
Time Frame: Weeks 24 and 48
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Then Dupilumab | Dupilumab
Number analyzed (Participants) | 20 | 40
score on a scale
  Week 24 | 4.29 (9.14) | 2.06 (8.49)
  Week 48 | 22.6 (35.42) | 8.13 (27.65)

9. Secondary Outcome: Eyelash/Eyebrow Assessment Score Weeks 12, 24, 36, and 48 Compared to Baseline
Description: Change in eyelash and eyebrow scores at Weeks 12, 24, 36, and 48 compared to baseline. The Eyelash/Eyebrow Assessment score based on a 5-point scale, ranging from 0 (none) to 4 (very prominent eyelashes/eyebrows).
Time Frame: Weeks 12, 24, 36, and 48
Population: One participant had missing eyelash data because of artificial eyelashes (glued on her real eyelashes).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Then Dupilumab | Dupilumab
Number analyzed (Participants) | 20 | 40
score on a scale
  Eyelash Week 12: number analyzed (Participants) | 19 | 40
  Eyelash Week 12 | 0 (0.37) | 0.07 (0.24)
  Eyelash Week 24: number analyzed (Participants) | 19 | 40
  Eyelash Week 24 | 0.37 (0.34) | 0.04 (0.24)
  Eyelash Week 36: number analyzed (Participants) | 19 | 40
  Eyelash Week 36 | -0.15 (0.37) | -0.06 (0.27)
  Eyelash Week 48: number analyzed (Participants) | 19 | 40
  Eyelash Week 48 | -0.17 (0.35) | 0.05 (0.26)
  Eyebrow Week 12 | 0.09 (0.37) | 0.21 (0.25)
  Eyebrow Week 24 | 0.27 (0.34) | 0.19 (0.24)
  Eyebrow Week 36 | -0.2 (0.34) | 0.17 (0.24)
  Eyebrow Week 48 | -0.03 (0.35) | 0.09 (0.25)

10. Secondary Outcome: Change in EASI Scores From Baseline at Week 24 and 48
Description: Change from baseline in Eczema Area and Severity Index (EASI) at Weeks 24 and 48. EASI scores range from 0 (no symptoms) to 72 (severe eczema) with lower score indicating better health outcomes/less eczema.
Time Frame: Weeks 24 and 48
Population: Data for only those participants with eczema.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Then Dupilumab | Dupilumab
Number analyzed (Participants) | 2 | 3
score on a scale
  Week 24 | -1.45 (3.61) | 10.6 (3.64)
  Week 48 | 23.9 (10.61) | 10.53 (3.75)

11. Secondary Outcome: Number of Adverse Events
Description: Safety profile of dupilumab in subjects with AA by reported adverse effects, physical examinations and laboratory parameters
Time Frame: 48 weeks
Measure: Number; unit: events
Arm/Group | Placebo Then Dupilumab | Dupilumab
Number analyzed (Participants) | 20 | 40
events | 24 | 9

ADVERSE EVENTS:
Time Frame: 48 weeks
Groups:
- Placebo: Matching placebo in prefilled syringes identical to the dupilumab syringes. 24 weeks of Placebo
- Dupilumab: Matching placebo in prefilled syringes identical to the dupilumab syringes. After 24 weeks of Placebo, an initial dose of 600 mg Dupilumab (two 300 mg subcutaneous injections), followed by an open-label period in which 300 mg given every other week. A total of 24 Dupilumab doses.
Arm/Group | Placebo | Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/40
Other Adverse Events (participants affected / at risk) | 4/20 | 22/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Dupilumab (N=40)
Bladder Cancer (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Dupilumab (N=40)
Injection site reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eosinophilic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gastrointestinal symptoms (Gastrointestinal disorders) | 1 (1) | 3 (3)
Other orthopedic injuries/procedures (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Bladder malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Facial rash (Infections and infestations) | 0 (0) | 1 (1)
Conjuctivitis (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 6 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT03359356/Prot_SAP_000.pdf